CLINICAL TRIAL: NCT07311343
Title: Oral Hygiene and Prophylactic Antibiotics to Prevent Intracerebral Hemorrhage Associated Pneumonia
Acronym: OCEAN
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, guojunping, Associate Chief Nurse, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KY2025-105-03
Record Dates: First submitted 2025-11-26; First posted 2025-12-30 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Hemorrhage; Pneumonia
Keywords: Cerebral hemorrhage; Stroke Associated Pneumonia; oral care; prophylactic antibiotics; effectiveness
MeSH Terms: conditions — Hemorrhage; Pneumonia; Cerebral Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- enhanced oral care combined with prophylactic antibiotics (Active Comparator): After randomization, immediate intensive oral hygiene treatment (chlorhexidine 20ml, three times a day) combined with antibiotics (ceftazidime 1g, every 8 hours) was given on the basis of conventional standard treatment, and the treatment course was 3 days.
  Interventions: Biological: wether apply enhanced oral care combined with prophylactic antibiotics
- conventional standard treatment combined with conventional oral care (Experimental): Conventional standard treatment combined with routine oral care (20 ml of normal saline twice a day), and detailed records were made of the specific measures of the patients' oral care, including the selection of the cleaning solution and the frequency.
  Interventions: Biological: wether apply enhanced oral care combined with prophylactic antibiotics

INTERVENTIONS:
Biological: wether apply enhanced oral care combined with prophylactic antibiotics — Intervention group: After randomization, immediate intensive oral hygiene treatment (chlorhexidine 20 ml, three times a day) combined with antibiotics (ceftazidime 1 g, every 8 hours) was administered on the basis of the conventional standard treatment, and the treatment lasted for 3 days; Control group: Conventional standard treatment combined with routine oral care (normal saline 20 ml, twice a day), and detailed records were made of the specific measures of patient oral care, including the selection of cleaning solution and frequency.

SUMMARY:
Project Name:

Randomized Controlled Clinical Study on oral hygiene and prophylactic antibiotics to prevent Intracerebral Hemorrhage associated pneumonia

Research Objectives:

To evaluate the effectiveness, safety and health economics value of enhanced oral hygiene combined with antibiotics in preventing post-cerebral hemorrhage pneumonia.

1. To clarify the effectiveness of enhanced oral hygiene combined with antibiotics in preventing post-cerebral hemorrhage pneumonia.
2. To clarify the safety of enhanced oral hygiene combined with antibiotics in preventing post-cerebral hemorrhage pneumonia.
3. To clarify the health economics value of low-intensity enhanced oral hygiene combined with antibiotics in preventing post-cerebral hemorrhage pneumonia.

Research Design:

Research Type: Multicenter, Randomized, Controlled, Open Label, Blinded Endpoint Research Design Research Hypothesis: Intensive oral hygiene combined with antibiotic treatment is beneficial in reducing the incidence of pulmonary infections related to cerebral hemorrhage.

DETAILED DESCRIPTION:
Research Background:

The era of evidence-based medicine has been entered. For acute ischemic stroke within the 4.5-hour time window, intravenous thrombolysis, mechanical thrombectomy within 24 hours of onset, and stroke units all have clear evidence-based medical support for their intervention methods. However, for cerebral hemorrhage, which has higher disability and mortality rates, treatment methods currently lack evidence-based medical support, with management more often being supportive. In this context, exploring new targets, methods, and strategies to improve the prognosis of cerebrovascular diseases has become a hot topic in global research.

Stroke-associated pneumonia (SAP) is one of the most common complications after stroke. Substantial evidence shows that the occurrence of SAP not only increases patient length of hospital stay and medical expenses but also significantly elevates the risk of death and severe disability post-stroke. Based on data from the China National Stroke Registry (CNSR), the composition and distribution of various complications after cerebral infarction and cerebral hemorrhage in Chinese patients were first systematically reported. Among them, SAP is the most common complication for both major stroke subtypes: cerebral infarction and cerebral hemorrhage. Concurrently, it was also found that SAP not only increases the risk of adverse stroke prognosis but is also an important risk factor for the increase of various non-pneumonia complications. For example, in the sub-cohort of acute cerebral infarction patients (N=14,702), the occurrence of SAP increased the risk of gastrointestinal bleeding by 8-fold (adjusted OR=8.35; 95% CI=6.27-11.1; P<0.001), pressure ulcers by 5-fold (OR=5.31; 95% CI=3.39-8.31; P<0.001), deep vein thrombosis by 4-fold (OR=4.27; 95% CI=2.41-7.59; P<0.001), symptomatic epilepsy by 4-fold (OR=3.96; 95% CI=2.67-5.88; P<0.001), urinary tract infection by 3-fold (OR=3.34; 95% CI=2.73-4.10; P<0.001), atrial fibrillation by 3-fold (OR=3.17; 95% CI=2.58-3.90; P<0.001), and stroke recurrence by 2-fold (OR=2.65; 95% CI=2.07-3.40; P<0.001).

The same phenomenon was also confirmed in the cerebral hemorrhage cohort (N=5,221). The effective prevention and control of SAP will become a new target for improving stroke prognosis, as clearly reflected in multiple domestic and international expert consensuses and guidelines on SAP.

Similar related studies have been conducted abroad. In 2015, the UK STROKE-INF study, for patients hospitalized within 48 hours after stroke onset, administered prophylactic antibiotics for 7 days plus standard stroke ward care or standard stroke ward care alone, finally including 1,217 patients from 37 units (615 in the antibiotic group, 602 in the control group). No difference was found in the diagnosis of post-stroke pneumonia between the two groups (101 of 615 patients [16%] in the antibiotic treatment group vs. 91 of 602 patients [15%] in the non-antibiotic treatment group; adjusted OR = 1.01 [95% CI 0.61-1.68], p = 0.957). In 2015, the Dutch PASS study randomly assigned acute stroke patients in a 1:1 ratio to an antibiotic treatment group (ceftriaxone) or a non-antibiotic treatment group (control) within 24 hours after onset. The control group received standardized stroke treatment; the ceftriaxone group received standardized treatment plus intravenous application of 2g ceftriaxone once daily for 4 days. Finally, 2,538 patients were included for treatment analysis (ceftriaxone group: 1,268; control group: 1,270). The study results showed that prophylactic use of ceftriaxone was safe, mainly manifested by a significantly lower incidence of urinary tract infections in the ceftriaxone group, with no significant difference in the incidence of infections at other sites between the two groups. Prophylactic ceftriaxone did not affect the distribution of 3-month modified Rankin Scale (mRS) scores (OR = 0.95 [95% CI 0.81-1.09], p = 0.46). Both these trials yielded negative results. This study aims to explore the relationship between the preventive use of antibiotics combined with oral care and the incidence of SAP in the Chinese population.

Research Objectives:

To clarify the effectiveness of enhanced oral hygiene combined with antibiotics in preventing pneumonia after cerebral hemorrhage.

To clarify the safety of enhanced oral hygiene combined with antibiotics in preventing pneumonia after cerebral hemorrhage.

To clarify the health economics value of enhanced oral hygiene combined with antibiotics in preventing pneumonia after cerebral hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old;
2. Spontaneous intracerebral hemorrhage;
3. Supratentorial intracerebral hemorrhage (ICH);
4. Hematoma volume < 30 ml (calculated by ABC/2 method);
5. Glasgow Coma Scale score ≥ 9 at randomization;
6. Time from onset to randomization ≤ 72 hours;
7. Spontaneous intracerebral hemorrhage-associated pneumonia score (ICH-APS) ≥ 8;
8. Informed consent from the patient and/or their family.

Exclusion Criteria:

1. Secondary intracerebral hemorrhage, such as that resulting from cerebral aneurysms, cerebral arteriovenous malformations, brain tumors, cerebral venous system thrombosis, antithrombotic therapy (antiplatelet, anticoagulant therapy, etc.), hemorrhagic transformation after cerebral infarction, hematological diseases, etc.
2. The patient's clinical symptoms and signs suggest signs of brain herniation, such as progressive decline in consciousness level, weakened or absent pupillary light reflex.
3. Obvious signs of pneumonia already exist, such as fever, persistent cough or yellow purulent sputum, and imaging examinations (chest X-ray or chest CT) suggest signs of pneumonia; two consecutive measurements of body temperature ≥ 37.5℃, or one measurement of body temperature ≥ 38.0℃.
4. A history of severe cardiovascular disease, meeting any of the following: 1) Heart failure (New York Heart Association functional class ≥ III); 2) Unstable angina within 3 months; 3) Any supraventricular or ventricular arrhythmia requiring treatment; 4) Prolonged QTc interval considered clinically significant by the investigator (reference range: > 450ms for men, > 470ms for women) (Note: QTc interval must be calculated according to Fridericia's formula); 5) Complete atrioventricular block and left or right bundle branch block requiring treatment; 6) Acute myocardial infarction or interventional treatment within 1 month; high-risk patients with chronic arrhythmia, such as sick sinus syndrome, second or third-degree atrioventricular block, bradycardia-related syncope without pacemaker installation, etc.
5. Diagnosed with severe active liver disease, such as acute hepatitis, chronic active hepatitis, liver cirrhosis, etc.; or ALT or AST > 3 times the upper limit of normal.
6. Severe renal insufficiency: such as patients undergoing dialysis, or diagnosed with severe active kidney disease, etc., or creatinine clearance rate < 50 mL/min.
7. Other severe diseases that lead to an expected lifespan of less than 1 year.
8. Patients scheduled for surgical intervention before the first administration, including but not limited to hematoma evacuation (including minimally invasive and conventional surgery), decompressive craniectomy, hematoma aspiration, and external ventricular drainage.
9. Patients unable to understand the research procedures and/or complete follow-up due to mental illness, cognitive impairment, emotional disorders, etc.
10. Pregnant or lactating women.
11. Participation in other clinical studies within 3 months or currently participating in other clinical studies.
12. Known allergy to cephalosporins, penicillins, or chlorhexidine compound mouthwash.

    -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2026-01-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
The occurrence of pneumonia related to cerebral hemorrhage | From enrollment to the 10th day after randomization or at the time of discharge
  The occurrence of pneumonia related to cerebral hemorrhage

SECONDARY OUTCOMES:
urinary tract infection or other systemic infection | From enrollment to the 10th day after randomization or at discharge
  urinary tract infection or other systemic infection
Improvement in neurological dysfunction (NIHSS10d-NIHSS group) | From enrollment to the 10th day after randomization or at discharge
  This study used the difference between the NIH Stroke Scale (NIHSS, 0-42) score on the 10th day after randomization or at discharge and the NIHSS score (0-42) at the time of enrollment to represent the change in neurological dysfunction (NIHSS10d-NIHSS group). The smaller the difference, or even a negative value, the better the improvement in neurological dysfunction. Conversely, the larger the difference, the worse the improvement.
Length of hospital stay | From hospital admission until discharge (anticipated average 7-10 days)
  The period from the patient's admission to the patient's discharge.It is the date of discharge minus the date of admission
direct medical expenses during hospitalization | From hospital admission until discharge (anticipated average 7-10 days)
  The direct expenses incurred by the patient during the hospitalization period.
Modified Rankin Scale score | From enrollment to the 90 days ± 7 days after randomization
  This study used the Modified Rankin Scale (mRS，0-6) score at 90 ± 7 days after randomization to reflect the long-term prognosis of the patients. The higher the score, the worse the prognosis. Conversely, the lower the score, the better the prognosis.

CONTACTS AND LOCATIONS:
Overall Officials: Junping Guo, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Westendorp WF, Vermeij JD, Zock E, Hooijenga IJ, Kruyt ND, Bosboom HJ, Kwa VI, Weisfelt M, Remmers MJ, ten Houten R, Schreuder AH, Vermeer SE, van Dijk EJ, Dippel DW, Dijkgraaf MG, Spanjaard L, Vermeulen M, van der Poll T, Prins JM, Vermeij FH, Roos YB, Kleyweg RP, Kerkhoff H, Brouwer MC, Zwinderman AH, van de Beek D, Nederkoorn PJ; PASS investigators. The Preventive Antibiotics in Stroke Study (PASS): a pragmatic randomised open-label masked endpoint clinical trial. Lancet. 2015 Apr 18;385(9977):1519-26. doi: 10.1016/S0140-6736(14)62456-9. Epub 2015 Jan 20. PMID 25612858
- [Background] Kalra L, Irshad S, Hodsoll J, Simpson M, Gulliford M, Smithard D, Patel A, Rebollo-Mesa I; STROKE-INF Investigators. Prophylactic antibiotics after acute stroke for reducing pneumonia in patients with dysphagia (STROKE-INF): a prospective, cluster-randomised, open-label, masked endpoint, controlled clinical trial. Lancet. 2015 Nov 7;386(10006):1835-44. doi: 10.1016/S0140-6736(15)00126-9. Epub 2015 Sep 3. PMID 26343840
- [Background] Vernino S, Brown RD Jr, Sejvar JJ, Sicks JD, Petty GW, O'Fallon WM. Cause-specific mortality after first cerebral infarction: a population-based study. Stroke. 2003 Aug;34(8):1828-32. doi: 10.1161/01.STR.0000080534.98416.A0. Epub 2003 Jul 10. PMID 12855836
- [Background] Saposnik G, Hill MD, O'Donnell M, Fang J, Hachinski V, Kapral MK; Registry of the Canadian Stroke Network for the Stroke Outcome Research Canada (SORCan) Working Group. Variables associated with 7-day, 30-day, and 1-year fatality after ischemic stroke. Stroke. 2008 Aug;39(8):2318-24. doi: 10.1161/STROKEAHA.107.510362. Epub 2008 Jun 19. PMID 18566303
- [Background] Katzan IL, Dawson NV, Thomas CL, Votruba ME, Cebul RD. The cost of pneumonia after acute stroke. Neurology. 2007 May 29;68(22):1938-43. doi: 10.1212/01.wnl.0000263187.08969.45. PMID 17536051
- [Background] Ingeman A, Andersen G, Hundborg HH, Svendsen ML, Johnsen SP. In-hospital medical complications, length of stay, and mortality among stroke unit patients. Stroke. 2011 Nov;42(11):3214-8. doi: 10.1161/STROKEAHA.110.610881. Epub 2011 Aug 25. PMID 21868737
- [Background] Ji R, Wang D, Shen H, Pan Y, Liu G, Wang P, Wang Y, Li H, Wang Y; China National Stroke Registry (CNSR) Investigators. Interrelationship among common medical complications after acute stroke: pneumonia plays an important role. Stroke. 2013 Dec;44(12):3436-44. doi: 10.1161/STROKEAHA.113.001931. Epub 2013 Oct 31. PMID 24178914
- [Background] Kumar S, Selim MH, Caplan LR. Medical complications after stroke. Lancet Neurol. 2010 Jan;9(1):105-18. doi: 10.1016/S1474-4422(09)70266-2. PMID 20083041
- [Background] Badve MS, Zhou Z, van de Beek D, Anderson CS, Hackett ML. Frequency of post-stroke pneumonia: Systematic review and meta-analysis of observational studies. Int J Stroke. 2019 Feb;14(2):125-136. doi: 10.1177/1747493018806196. Epub 2018 Oct 22. PMID 30346258
- [Background] Steiner T, Al-Shahi Salman R, Beer R, Christensen H, Cordonnier C, Csiba L, Forsting M, Harnof S, Klijn CJ, Krieger D, Mendelow AD, Molina C, Montaner J, Overgaard K, Petersson J, Roine RO, Schmutzhard E, Schwerdtfeger K, Stapf C, Tatlisumak T, Thomas BM, Toni D, Unterberg A, Wagner M; European Stroke Organisation. European Stroke Organisation (ESO) guidelines for the management of spontaneous intracerebral hemorrhage. Int J Stroke. 2014 Oct;9(7):840-55. doi: 10.1111/ijs.12309. Epub 2014 Aug 24. PMID 25156220
- [Background] Hemphill JC 3rd, Greenberg SM, Anderson CS, Becker K, Bendok BR, Cushman M, Fung GL, Goldstein JN, Macdonald RL, Mitchell PH, Scott PA, Selim MH, Woo D; American Heart Association Stroke Council; Council on Cardiovascular and Stroke Nursing; Council on Clinical Cardiology. Guidelines for the Management of Spontaneous Intracerebral Hemorrhage: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2015 Jul;46(7):2032-60. doi: 10.1161/STR.0000000000000069. Epub 2015 May 28. PMID 26022637
- [Background] Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL. Guidelines for the Early Management of Patients With Acute Ischemic Stroke: 2019 Update to the 2018 Guidelines for the Early Management of Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2019 Dec;50(12):e344-e418. doi: 10.1161/STR.0000000000000211. Epub 2019 Oct 30. PMID 31662037
- [Background] Wang W, Jiang B, Sun H, Ru X, Sun D, Wang L, Wang L, Jiang Y, Li Y, Wang Y, Chen Z, Wu S, Zhang Y, Wang D, Wang Y, Feigin VL; NESS-China Investigators. Prevalence, Incidence, and Mortality of Stroke in China: Results from a Nationwide Population-Based Survey of 480 687 Adults. Circulation. 2017 Feb 21;135(8):759-771. doi: 10.1161/CIRCULATIONAHA.116.025250. Epub 2017 Jan 4. PMID 28052979
- [Background] GBD 2016 Neurology Collaborators. Global, regional, and national burden of neurological disorders, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2019 May;18(5):459-480. doi: 10.1016/S1474-4422(18)30499-X. Epub 2019 Mar 14. PMID 30879893
- [Background] Feigin VL, Roth GA, Naghavi M, Parmar P, Krishnamurthi R, Chugh S, Mensah GA, Norrving B, Shiue I, Ng M, Estep K, Cercy K, Murray CJL, Forouzanfar MH; Global Burden of Diseases, Injuries and Risk Factors Study 2013 and Stroke Experts Writing Group. Global burden of stroke and risk factors in 188 countries, during 1990-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet Neurol. 2016 Aug;15(9):913-924. doi: 10.1016/S1474-4422(16)30073-4. Epub 2016 Jun 9. PMID 27291521
- [Background] GBD 2015 DALYs and HALE Collaborators. Global, regional, and national disability-adjusted life-years (DALYs) for 315 diseases and injuries and healthy life expectancy (HALE), 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1603-1658. doi: 10.1016/S0140-6736(16)31460-X. PMID 27733283
- [Background] Wu S, Wu B, Liu M, Chen Z, Wang W, Anderson CS, Sandercock P, Wang Y, Huang Y, Cui L, Pu C, Jia J, Zhang T, Liu X, Zhang S, Xie P, Fan D, Ji X, Wong KL, Wang L; China Stroke Study Collaboration. Stroke in China: advances and challenges in epidemiology, prevention, and management. Lancet Neurol. 2019 Apr;18(4):394-405. doi: 10.1016/S1474-4422(18)30500-3. PMID 30878104
- [Background] Virani SS, Alonso A, Benjamin EJ, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Shay CM, Spartano NL, Stokes A, Tirschwell DL, VanWagner LB, Tsao CW; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2020 Update: A Report From the American Heart Association. Circulation. 2020 Mar 3;141(9):e139-e596. doi: 10.1161/CIR.0000000000000757. Epub 2020 Jan 29. PMID 31992061